CLINICAL TRIAL: NCT07266090
Title: A Multicenter,Open-label,Single Arm,Multiple-dose Study to Evaluate the Safety,Tolerability,Pharmacokinetics and Pharmacodynamics of Cenerimod in Adult Chinese Participants With Moderate-to-severe Systemic Lupus Erythematosus (SLE) on Top of Background Therapy
Brief Title: A Study to Evaluate the Safety,Tolerability,Pharmacokinetics and Pharmacodynamics of Cenerimod in Adult Chinese Participants With Moderate-to-severe Systemic Lupus Erythematosus (SLE)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Viatris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID-064A204
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: SLE - Systemic Lupus Erythematosus
Keywords: cenerimod; ACT-334441; safety; tolerability; pharmacokinetics; pharmacodynamics; Chinese participants
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — cenerimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cenerimod (Experimental): cenerimod 4 mg once daily
  Interventions: Drug: cenerimod 4 mg

INTERVENTIONS:
Drug: cenerimod 4 mg — cenerimod 4 mg once daily for 12 months

SUMMARY:
The goal of this clinical trial is to learn about the safety, how the body processes the drug, and its effects of a drug called cenerimod in adult Chinese participants (aged 18-75) with moderate to severe Systemic Lupus Erythematosus (SLE) who are already receiving standard background therapy.

The main questions it aims to answer are:

* What is the safety and tolerability of a daily 4 mg dose of cenerimod in Chinese participants with SLE?
* How is cenerimod processed by the body (pharmacokinetics) in this population?
* What is the effect of cenerimod on the level of lymphocytes in the blood (pharmacodynamics)? This is a single-arm study without a comparison group.

Participants will:

* Take one 4 mg cenerimod tablet by mouth once daily for up to 12 months.
* Continue their stable, pre-existing background SLE medications throughout the study.
* Attend regular clinic visits over a period of up to 22 months for tests and check-ups, including blood draws, heart monitoring (12-lead electrocardiogram), vital signs(blood pressure),and physical examinations.
* Undergo a final safety follow-up 6 months after their last dose of the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated ICF prior to any study-mandated procedure.
2. Male and female Chinese participants aged from 18 to 75 years old (inclusive) at the time of signing the ICF.
3. Diagnosis of SLE made at least 6 months prior to Screening, according to 2019 European League Against Rheumatism / American College of Rheumatology Criteria.
4. An mSLEDAI-2K score ≥ 6 and clinical mSLEDAI-2K score ≥ 4 with at least 2 points for musculoskeletal or mucocutaneous manifestations (i.e., myositis, arthritis, rash, alopecia, mucosal ulcers).

   Note: The mSLEDAI-2K score does not include "leukopenia". The clinical mSLEDAI-2K is the mSLEDAI-2K assessment score without the inclusion of points attributable to hematuria, proteinuria, pyuria, urinary casts, low complement, increased DNA binding, and thrombocytopenia.
5. PGA score ≥ 1.0 on a 0 to 3 VAS.
6. Currently treated with one or more of the following SLE background medications:

   * Antimalarials: (≤ 400 mg/day hydroxychloroquine, ≤ 500 mg/day chloroquine, ≤ 100 mg/day quinacrine),
   * Mycophenolate mofetil (≤ 2 g/day) / mycophenolic acid (≤ 1.44 g/day),
   * Azathioprine (≤ 2 mg/kg/day),
   * Methotrexate (≤ 25 mg/week),
   * Oral corticosteroid(s) (OCS):

     * If OCS is the only SLE background medication:

       ≥ 7.5 mg/day and ≤ 30 mg/day prednisone or equivalent.
     * If OCS is not the only SLE background medication:

       * 30 mg/day prednisone or equivalent.
   * Belimumab (≤ 10 mg/kg every 4 weeks intravenously [i.v.] or ≤ 200 mg/week subcutaneously [s.c.]).
   * Telitacicept (≤ 240 mg/week subcutaneously). Treatment with antimalarials, mycophenolate mofetil, mycophenolic acid, azathioprine, methotrexate, belimumab, or telitacicept must have been started at least 90 days prior to Screening.

   Treatment with OCS must have been started at least 30 days prior to Screening.
7. For women of childbearing potential (WoCBP):

   * Negative serum pregnancy test at Screening.
   * Agreement to undertake monthly urine pregnancy tests from Day 1 up to 6 months after study treatment discontinuation.
   * Agreement to use a highly effective method of contraception from Screening (Visit 1) up to 6 months after study treatment discontinuation.
8. On Day 1 before dosing,A clinical mSLEDAI-2K score ≥ 4 with at least 2 points for musculoskeletal or mucocutaneous manifestations (i.e., myositis, arthritis, rash, alopecia, mucosal ulcers).
9. On Day 1 before dosing,PGA score ≥ 1.0 on a 0 to 3 VAS.
10. On Day 1 before dosing,Presence of at least one of the following biomarkers of serological evidence of active SLE (in a Screening sample as measured by central laboratory):

    * Anti-dsDNA antibodies elevated above normal.
    * Antinuclear antibodies (ANA) with a titer of at least 1:160.
    * Anti-Smith (anti-Sm) antibody elevated above normal.
11. On Day 1 before dosing,Currently treated with one or more of the following SLE background medications that must be stable for at least 30 days prior to Day 1 (except OCS, which must be stable for at least 15 days prior to Day 1):

    * Antimalarials (≤ 400 mg/day hydroxychloroquine, ≤ 500 mg/day chloroquine, ≤ 100 mg/day quinacrine),
    * Mycophenolate mofetil (≤ 2 g/day) / mycophenolic acid (≤ 1.44 g/day),
    * Azathioprine (≤ 2 mg/kg/day),
    * Methotrexate (≤ 25 mg/week),
    * OCS:

      * If OCS is the only SLE background medication:

        * 7.5 mg/day and ≤ 30 mg/day prednisone or equivalent.
      * If OCS is not the only SLE background medication:

        * 30 mg/day prednisone or equivalent.
    * Belimumab (≤ 10 mg/kg every 4 weeks i.v. or

      ≤ 200 mg/week s.c.);
    * Telitacicept (≤ 240 mg/week subcutaneously).
12. On Day 1 before dosing,WoCBP must have a negative urine pregnancy test.

Exclusion Criteria:

1. Pregnant, planning to be become pregnant up to 6 months after the last dose of cenerimod in this study, or lactating women.
2. Active severe SLE-driven renal disease (within 90 days prior to Screening or during Screening) where, in the judgment of the investigator, protocol-specified SLE background therapy is insufficient and the use of a more aggressive therapeutic approach or other treatments not permitted in the protocol is indicated.
3. Urine protein/creatinine ratio> 3000 mg/g (i.e., > 339.45 mg/mmol) at Screening assessment based on central assessment.
4. Severe active central nervous system lupus or active severe or unstable neuropsychiatric SLE including but not limited to: aseptic meningitis; cerebral vasculitis; myelopathy; demyelination syndromes (ascending, transverse, acute inflammatory demyelinating polyradiculopathy); acute confusional state; impaired level of consciousness; psychosis; acute stroke or stroke syndrome; cranial neuropathy; status epilepticus; cerebellar ataxia; or mononeuritis multiplex:

   * That would make the participant unable to fully understand the ICF. or
   * Where, in the opinion of the investigator/delegate, protocol-specified standard of care is insufficient and the use of a more aggressive therapeutic approach, such as adding i.v. cyclophosphamide and/or high dose i.v. pulse corticosteroid (CS) therapy or other treatments not permitted in the protocol is indicated.
5. Severe forms of vasculitis (e.g., retinal vasculitis, coronary vasculitis, pulmonary vasculitis, mesenteric vasculitis) requiring systemic immunosuppressive treatment within 90 days prior to Screening or during Screening.
6. A diagnosis of mixed connective tissue disease or any history of overlap syndromes of SLE with psoriasis, rheumatoid arthritis, erosive arthritis, scleroderma, autoimmune hepatitis, or uncontrolled autoimmune thyroid disease.
7. History or presence of Mobitz type II or third-degree atrioventricular block, sick sinus syndrome, symptomatic bradycardia, or syncope associated with cardiac disorders.
8. Participants who experienced myocardial infarction, unstable angina pectoris, stroke, transient ischemic attack, vascular thrombosis, decompensated heart failure requiring hospitalization, or heart failure defined by the New York Heart Association Class III/IV (see Appendix 14) within 6 months prior to Screening.
9. Resting HR < 50 beats per minute as measured by the 12-lead ECG at Screening or at Day 1 prior to study treatment administration.
10. An elevated QTcF interval of > 470 ms (females) / > 450 ms (males) at Screening or at Day 1 prior to study treatment administration.
11. History or presence of severe respiratory disease or pulmonary fibrosis, based on medical history, lung function, and chest X-ray (or CT scan as per local guidelines), performed at Screening or within 6 months prior to Screening.
12. History of clinically relevant bronchial asthma or chronic obstructive pulmonary disease that has required treatment with oral or parenteral CS for more than a total of 2 weeks within the last 6 months prior to Screening.
13. Have had household contact with a person with active Tuberculosis (TB) and did not receive appropriate and documented prophylaxis for TB.
14. Have evidence of active TB or latent TB

    1. Active TB: Have evidence of active TB, defined in this study as the following:

       * Medical history, clinical features, and abnormal chest X- ray at Screening indicating the presence of TB.
       * IFN gamma release assay (IGRA): participants are excluded from the study if the test is not negative and there is clinical evidence of active TB.

       Exception 1: participants with a history of active TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, have no clinical features of active TB, and have a Screening chest X-ray with no evidence of active TB may be enrolled if other entry criteria met. Such participants would not be required to undergo the IGRA test, but must have a chest X- ray at Screening (i.e., chest imaging performed within the past 6 months will not be accepted).
    2. Latent TB: Have evidence of untreated/inadequately or inappropriately treated latent TB, defined in this study as the following:

       * An IGRA test which is not negative, no clinical features consistent with active TB, and a chest X-ray with no evidence of active TB at Screening;
       * If the IGRA test results are positive, the participant will be considered to have latent TB. If the test is not negative, the test may be repeated once within approximately 2 weeks of the initial value. If the repeat test results are again not negative, the participant will be considered to have latent TB (for purposes of this study).

    Exception 2: participants with a history of latent TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, have no clinical features of active TB, and have a Screening chest X-ray with no evidence of active TB may be enrolled if other entry criteria met. Such participants would not be required to undergo the IGRA test, but must have a chest X- ray at Screening (i.e., chest imaging performed within the past 6 months will not be accepted).
15. Ongoing bacterial, viral, parasitic, or fungal infection that is of clinical concern according to the investigator or any of the following:

    * Clinically significant chronic infection (e.g., osteomyelitis, bronchiectasis, etc.) within 8 weeks prior to Screening (chronic nail infections are allowed).
    * Any infection requiring hospitalization or treatment with i.v. anti-infectives not completed at least 4 weeks prior to Screening.
16. Positive results for serological markers for hepatitis A, B, C, and E indicating acute or chronic infection:

    * Anti-hepatitis A virus (HAV) immunoglobulin M (IgM).
    * Hepatitis B surface antigen.
    * Anti-hepatitis C virus (HCV) IgG or IgM (if positive IgM and/or IgG, to be confirmed by HCV-RNA polymerase chain reaction assessment, and if this assessment is negative, participant can be enrolled).
    * Anti-hepatitis E virus (HEV) IgG or IgM (if positive IgM and/or IgG, to be confirmed by HEV-RNA polymerase chain reaction, and if this assessment is negative, participant can be enrolled).
17. Participants who have congenital or acquired severe immunodeficiency or known human immunodeficiency virus (HIV) infection or positive HIV testing.
18. Negative IgG antibody test for varicella-zoster virus.
19. History or presence of malignancy (except for surgically excised and non-recurrent cutaneous basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma), lymphoproliferative disease, or history of total lymphoid irradiation within 10 years prior to Screening.
20. History or presence of homologous (allogenic) bone marrow or solid organ transplantation.
21. Presence of macular edema or active uveitis detected by optical coherence tomography (OCT) during Screening.
22. Documented poorly controlled diabetes mellitus (i.e., glycated hemoglobin > 8.0% at Screening as reported by the central laboratory or unstable blood sugar control/treatment adherence as per investigator's judgment) or diabetes mellitus complicated with organ involvement, such as diabetic nephropathy or retinopathy as assessed by investigator.
23. History of chronic liver or biliary disease (other than Gilbert's Syndrome) or participants with alanine aminotransferase or aspartate aminotransferase > 3 × upper limit of normal or total bilirubin > 1.5 ×upper limit of normal (unless in the context of known Gilbert's Syndrome).
24. Significant hematology abnormality at screening assessment:

    * Lymphocyte count < 500 /μL (0.5 × 10^9/L);
    * Hemoglobin < 7 g/dL;
    * White blood cell count < 2000/μL (2.0 × 10^9/L) or
    * Platelets < 25,000/μL (25 × 10^9/L).
25. Estimated glomerular filtration rate < 15 mL/min/1.73 m^2.
26. Treatment with the following medications within 15 days or 5 half-lives of the medication (whichever is longer) prior to Day 1:

    * β-blockers, diltiazem, verapamil, digoxin, digitoxin, or any other anti-arrhythmic or HR-lowering systemic therapy.
    * QT-prolonging drugs with known risk of torsade de pointes irrespective of indication.
27. Treatment with the following medications within 30 days or 5 half-lives of the medication (whichever is longer) prior to Day 1:

    * Cyclophosphamide, cyclosporine, voclosporin, tacrolimus, sirolimus, etc.
    * Pulse methylprednisolone.
    * Vaccination with live vaccines.
28. Intra-articular, intramuscular or i.v. CS within 6 weeks prior to Day 1.
29. Treatment with the following medications within 90 days or 5 half-lives of the medication (whichever is longer) prior to Day 1:

    * Leflunomide.
    * i.v. immunoglobulins.
30. Treatment with any investigational agent within 90 days or 5 half-lives of the drug (whichever is longer) prior to Day 1.
31. Treatment with B cell-depleting biological agents (e.g., rituximab or ocrelizumab) or biological immunosuppressive agents (e.g., anti-tumor necrosis factor, anti-interleukin- [IL]1, anti-IL-6 therapies), within 12 months prior to Day 1.
32. Treatment with anifrolumab within 6 months prior to Day 1.
33. Treatment with any of the following medications any time prior to Screening:

    * Alemtuzumab.
    * Sphingosine-1-phosphate (S1P) receptor modulators (e.g., fingolimod).
    * Participants previously randomized to cenerimod or placebo in any trial involving cenerimod.
34. Recent clinically significant drug or alcohol abuse as per investigator's judgment.
35. Known allergy to S1P receptor modulators or any of the cenerimod formulation excipients.
36. Any other clinically relevant medical condition that would put the participant at risk if participating in the study, or any other diseases that may confound the disease activity assessments.
37. Participants with body weight < 40 kg at Screening or Day 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2027-10-08 (Estimated); Study Completion 2027-10-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (AEs) | From first dose of study treatment up to 180 days after the last dose
  Treatment-emergent AEs are defined as any adverse event that occurs after the first dose of study treatment and up to 180 days after the last dose. This includes serious AEs (SAEs), AEs of special interest (AESIs), and AEs leading to permanent discontinuation of study treatment. AEs are coded using MedDRA and assessed by the investigator.
Occurrence of adverse events leading to permanent discontinuation of study treatment | From first dose of study treatment up to end of treatment,maximum duration of 12 months.
  Number of participants who permanently discontinue study treatment due to adverse events.
Change from baseline in vital signs (systolic and diastolic blood pressure) and body weight | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12
  Change in systolic blood pressure (SBP), diastolic blood pressure (DBP), and body weight from baseline to each post-baseline assessment. Measurements are performed in duplicate under standardized conditions.
Change from baseline in 12-lead electrocardiogram (ECG) parameters | Baseline, Month 1, Month 2, Month 3, Month 4,Month 5,Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12
  Change in heart rate (HR), PR interval, QRS interval, QTcB interval, and QTcF interval from baseline to each post-baseline assessment.ECG abnormalities are assessed based on pre-defined criteria.
Change from baseline in laboratory parameters | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12
  Change in hematology, blood chemistry, and urinalysis variables from baseline to each post-baseline assessment. Marked laboratory abnormalities are defined based on central laboratory reference ranges.
Cenerimod Plasma Concentration | Pre-dose (0h), and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, and 24 hours post-dose on Day 1; Pre-dose on Day 30 (Month 1); Pre-dose, and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, and 24 hours post-dose on Day 60 (Month 2); Pre-dose on Day 120 (Month 4); Pre-dose on Day 180
  Plasma concentrations of cenerimod are measured at multiple time points to characterize the pharmacokinetic profile. Concentrations are determined using a validated bioanalytical method (e.g., LC-MS/MS).
Maximum plasma concentration (Cmax) of cenerimod | Day 1 and Month 2
  Cmax is derived from plasma concentration-time profiles using non-compartmental analysis. Assessed during the first dosing interval on Day 1 and at steady state (Month 2).
Time to maximum plasma concentration (tmax) of cenerimod | Day 1 and Month 2
  tmax is derived from plasma concentration-time profiles using non-compartmental analysis. Assessed during the first dosing interval on Day 1 and at steady state (Month 2).
  Time Frame: Day 1 and Month 2
Area under the plasma concentration-time curve from time zero to 24 hours (AUC0-24) of cenerimod | Day 1
  AUC0-24 is derived during the first dosing interval on Day 1 using non-compartmental analysis.
Area under the plasma concentration-time curve over a dosing interval at steady state (AUCτ) of cenerimod | Month 2
  AUCτ is derived at steady state (Month 2) using non-compartmental analysis.
Accumulation index (AI) of cenerimod | Between Day 1 and Month 2
  AI is calculated as the ratio of AUC at steady state (Month 2) to AUC after the first dose (Day 1).
Change from baseline in total blood lymphocyte count | Baseline to Month 12
  Change in total blood lymphocyte count from baseline to each post-baseline assessment. This is a key pharmacodynamic marker for cenerimod.
Number of participants with treatment-emergent medically relevant ECG abnormalities | Baseline to Month 12
  Treatment-emergent medically relevant ECG abnormalities are defined as new or worsening abnormalities from baseline to each post-baseline assessment, as determined by central reading.
Number of participants with treatment-emergent marked laboratory abnormalities | Baseline to Month 12
  Treatment-emergent marked laboratory abnormalities are defined as new or worsening abnormalities in hematology, blood chemistry, or urinalysis from baseline to each post-baseline assessment, based on central laboratory criteria.

OTHER OUTCOMES:
Proportion of participants achieving Systemic Lupus Erythematosus Responder Index 4 (SRI-4) response | Baseline to Month 12
  SRI-4 response is defined as a reduction of ≥4 points in mSLEDAI-2K score, no new BILAG A organ domain score, no more than 1 new BILAG B organ domain score, and no worsening in Physician's Global Assessment (PGA) score (assessed on a 0-3 VAS).
Proportion of participants achieving response on modified Systemic Lupus Erythematosus Disease Activity Index 2000 (mSLEDAI-2K) | Baseline to Month 12
  Response is defined as a reduction in mSLEDAI-2K score from baseline. The mSLEDAI-2K assesses SLE disease activity without including "leukopenia" or laboratory items.
Proportion of participants achieving British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) response | Baseline to Month 12
  BICLA response is defined as improvement in all organ systems (reduction of all BILAG A scores to B/C/D and all B scores to C/D) with no worsening in other systems.
Proportion of participants achieving response on Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) | Baseline to Month 12
  CLASI response is defined as improvement in skin activity score. CLASI assesses cutaneous lupus manifestations.
Change from baseline in tender joint count | Baseline to Month 12
  Change in the number of tender joints from baseline to Month 12. Assessed by physical examination.
Change from baseline in oral corticosteroid (OCS) dosage | Baseline to Month 12
  Change in the dose of OCS (prednisone or equivalent) from baseline to Month 12. OCS dosage is managed per protocol-specified rules.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Peking Union Medical College Hospital, Beijing

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT07266090/Prot_SAP_000.pdf